CLINICAL TRIAL: NCT06502457
Title: Pain Management With Virtual Reality Hypnosis in Parturients in the Latency or Cervical Ripening Phase
Brief Title: Pain Management With Virtual Reality Hypnosis
Acronym: PreVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PI2024_843_0067
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hypnosis; Labor Pain; Virtual Reality; Labor Induction; Latent Period
Keywords: hypnosis; labor pain; virtual reality; labor induction; latent period
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Drug: painkiller
- hypnosis group (Experimental)
  Interventions: Other: hypnosis group

INTERVENTIONS:
Drug: painkiller — The control group will receive a painkiller adapted to the service protocol after the fetal heart rate has been recorded.
  Arms: control group
Other: hypnosis group — The hypnosis group will receive a hypnosis session after the fetal heart rate has been recorded. Automated measurement of blood pressure and maternal heart rate will take place during the session in order to objectively assess the impact of the session on the mother.
  Patients in the hypnosis group will then have access to the virtual reality headset on request throughout the latency or maturation phase, and will also be able to benefit from a painkiller in accordance with the service protocol if they so request.
  Arms: hypnosis group

SUMMARY:
The latency phase corresponds to the first phase of the first stage of labour, during which the parturient feels regular, rhythmic uterine contractions that are often painful, with or without changes of the cervix. This phase lasts an average of 8 hours for primiparous women, compared with 5 hours for multiparous women, and can last up to twenty hours in total.

Cervical ripening corresponds to the medical induction of regular, painful uterine contractions in order to obtain a favourable cervix for the induction of labour. Cervical ripening is carried out either medically (oral or local prostaglandins) or mechanically (double balloon dilatation) and accounts for 69.2% of labour inductions, which in turn account for 25.8% of births.

At Amiens-Picardie University Hospital, this maturation stage can last from a few hours to 2 days, depending on the service protocol.

What these two stages of childbirth have in common is that they are both painful, with very few analgesic drugs available that can be used without side-effects on the foetus during pregnancy.

In recent years, there has also been a growing demand from parturients for the use of non-medicinal therapies.

It therefore seems essential to provide parturients with as many effective non-drug methods as possible to manage their pain properly.

If virtual reality hypnosis sessions prove to be effective, they will provide better pain management for women in labour, reduce the use of morphine derivatives (with their attendant side-effects, particularly on the foetus), and above all meet the growing demand from women in labour for the most physiological possible support during childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Parturient over 18
* Parturient who speaks and understands French
* Parturient hospitalised prior to labour
* Membranes intact or ruptured
* Spontaneous or induced labour
* Parturient in latency phase
* Term ≥ 37SA
* END > 3
* Parturient requiring active pain management (medicinal or non-medicinal)
* Low-risk pregnancy

Exclusion Criteria:

* Parturient under legal protection
* Parturient with a hearing impairment
* Parturient with visual impairment
* Parturient with epilepsy
* Parturient with psychiatric problems
* Pathological pregnancy
* Parturient with chronic pain
* Parturient with addiction-related disorders
* Parturient allergic to paracetamol
* Parturient allergic to phloroglucinol
* Parturient allergic to codeine
* Parturient allergic to nalbuphine
* Parturient allergic to orozamudol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
pain intensity difference between the first analgesic procedure and 30min later | 30 minutes
  Assessment of PID (pain intensity difference) between the first analgesic procedure and 30min later.

SECONDARY OUTCOMES:
Average consumption of analgesics | 12 hours
  Average consumption of analgesics (morphine agonists and other analgesics) during the latency or maturation period.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No